CLINICAL TRIAL: NCT00984880
Title: Phase I, Single Centre, Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 After a Single Ascending Bolus Dose, and a Single Ascending Bolus Dose Followed by a Single Infusion Dose in Healthy Volunteers
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD3043
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0510C00002; Eudract number: 2008-005836-34
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Sedation; anaesthesia; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — AZD-3043

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intravenous solution given as a single ascending bolus dose
  Interventions: Drug: AZD3043
- 2 (Experimental): Intravenous solution given as a single ascending bolus dose followed by a single infusion
  Interventions: Drug: AZD3043

INTERVENTIONS:
Drug: AZD3043 — Intravenous solution given as bolus dose (part A) and as bolus dose followed by infusion (part B)

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AZD3043 following administration of single ascending bolus doses (Part A) and single ascending bolus doses followed by infusion (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suitable veins for cannulation or repeated venepuncture
* Pre-dose assessment judged without remarks by the investigator
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Abnormal vital signs, after 15 minutes supine rest, defined as any of the following:
* Systolic blood pressure >140 mm Hg
* Diastolic blood pressure >90 mm Hg
* Heart rate ≤45 or >85 beats per minute
* Lack of normal phenotype for BuChE (Butyrylcholinesterase)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-09; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Assessment of vital signs data, heart rate, ECG | The measure will be taken between -20 to 120 min relative to stop of administration of AZD3043
Respiratory signs data (SpO2, EtCO2, PaO2, blood gases, respiratory frequency and pattern, occurrence of apnoea) | The measure will be taken between -20 to 120 min relative to stop of administration of AZD3043

SECONDARY OUTCOMES:
PK parameters for AZD3043: Cmax (in part B: bolus Cmax and infusion Cmax), AUClast, AUC, lz, t½lz, CL, Vc, Vss, Vz, tmax, tlast and MRT arterial and venous plasma. | Part A: Arterial: Predose and continously up to 120 min after start of dosing. Part B: Arterial: Predose and continously up to 150 min after start of dosing. Venous: Predose and continously up to 24 h after start of dosing
PK parameters for the metabolite (THRX 108893): Cmax (in part B: bolus Cmax and infusion Cmax), AUClast, AUC, tmax, tlast, lz and t½lz in arterial and venous plasma. | Part A: Arterial: Predose and continously up to 120 min after start of dosing. Part B: Arterial: Predose and continously up to 150 min after start of dosing. Venous: Predose and continously up to 24 h after start of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Johan Wemer, Study Chair — AstraZeneca; Sigridur Kalman, Principal Investigator — Karolinska University Hospital; Stephen Kanes, Study Director — AstraZeneca
Locations (1):
- Research Site, Stockholm, Sweden

REFERENCES:
- [Derived] Norberg A, Koch P, Kanes SJ, Bjornsson MA, Barassin S, Ahlen K, Kalman S. A Bolus and Bolus Followed by Infusion Study of AZD3043, an Investigational Intravenous Drug for Sedation and Anesthesia: Safety and Pharmacodynamics in Healthy Male and Female Volunteers. Anesth Analg. 2015 Oct;121(4):894-903. doi: 10.1213/ANE.0000000000000804. PMID 26097986